CLINICAL TRIAL: NCT01213901
Title: Optimizing Insulin Absorption and Insulin Injection Technique in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Graydon Meneilly, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: H10-00462
Record Dates: First submitted 2010-09-29; First posted 2010-10-04 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Diabetes
Keywords: Insulin absorption; Insulin injection technique
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Each patient will receive 2 insulin injections in the abdomen: Once using a pinch method and once using a spread method.
  Injections will be given in a random order and the technician will be blinded to the injection.
  Each patient will evaluate the comfort of the injection by completing a visual analog scale.
  Interventions: Procedure: Lispro insulin

INTERVENTIONS:
Procedure: Lispro insulin — Each patient will receive 2 insulin injections in the abdomen: Once using a pinch method and once using a spread method.

SUMMARY:
To determine which anatomic site offers the most consistent (superior) absorption of insulin.

To determine the injection technique which allows the most consistent subcutaneous injection of insulin (to pinch or to spread).

Hypothesis:

Based on age-related changes in the amount of subcutaneous fat we anticipate that the absorption of insulin from various anatomical sites will differ.

Justification:

To date health care professionals have extrapolated data obtained from younger adults and applied the results to the elderly.

Objectives:

To determine the rate of insulin absorption from different anatomic sites in diabetic patients over the age of 70.

To determine the best practice for subcutaneous injection in older adults.

Research Method:

Measurement of serial glucose and insulin levels using 360 minute euglycemic clamp studies.

Statistical Analysis:

Paired t test, repeated measures ANOVA

DETAILED DESCRIPTION:
The study will consist of 5 visits to the UBC VITALiTY Research Centre. At the screening visit subjects will have the following information collected: height, weight, blood pressure, heart rate, BMI, medical history and concommitant medications. Approximately 15cc of blood will be drawn and analyzed for A1C, CBC with platelets, AST, ALT, alk phos, BUN, creatinine, fasting blood sugar.

The subjects will undergo 4 euglycemic clamp studies at least 30 days apart in random order. During one study subjects will receive the insulin injection in the abdomen using the pinch technique. In another study the subjects will receive the insulin injection using the spread technique. During a third study the subjects will receive the insulin injection in the deltiod area using the pinch technique. During a fourth study the subjects will receive the insulin injection in the deltoid using the spread technique. Subjects will be randomly assigned to the studies. After each injection the subject will complete a questionnaire to rate comfort of the injection.

Subjects will report to the Research Centre at 0700 having fasted since midnight the night before. An intravenous line with normal saline will be placed in one hand to facilitate blood drawing. This hand will be placed in a heated box. A second intravenous will be inserted in the arm for the infusion of glucose.

Prior to subcutaneous insulin injection, blood samples will be collected at -30, -15, and 0 minutes. At time 0 the subcutaneous injection of lispro insulin (0.1 u/kg)will be administered and the glucose infusion will be started. Glucose levels will be measured at the bedside every 5 min and insulin levels every 15 min from 0-360 min. Glucose infusion will be adjusted to maintain glucose levels at a constant level for the duration of the study, using the glucose clamp protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over the age of 70
* Type 2 diabetes
* Insulin naive - never have taken insulin with the exception of a short course during a hospitalization or illness
* A1C between .065-.085
* BMI between 25 and 35

Exclusion Criteria:

* hemoglobin below 130g/L (males) and below 120g/L (females)
* taking medications that are known to interfere with glucose metabolism: systemic corticosteroids, non selective beta blockers
* Impaired liver function as shown by but not limited to AST and/or ALT > 2 times the upper limit of normal
* impaired renal function as shown by but not limited to serum creatinine > 133micromoles/L (males) and 124 micromoles/L (female)
* participation in another clinical trial within the past 30 days

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Anatomic site, abdomen versus deltoid, that offers the most consistent(superior) absorption of insulin

SECONDARY OUTCOMES:
Injection technique which allows the most comfortable method of inserting the needle subcutaneously

CONTACTS AND LOCATIONS:
Overall Officials: Gale Tedder, Study Director — Vancouver Coastal Health Research Institute; Chris Lockhart, Study Director — Vancouver Coastal Health Research Institute; Lee Ann Trimble, Study Director — Vancouver Coastal Health Research Institute
Locations (1):
- Vitality Research Centre - Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Trimble LA, Meneilly GS. Optimizing insulin absorption and insulin injection technique in older adults. Diabetes Care. 2014 Jun;37(6):e127-8. doi: 10.2337/dc14-0086. No abstract available. PMID 24855165